CLINICAL TRIAL: NCT06293651
Title: an Open-Label, Phase 1/2a, First-in-Human Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of DA-4505 as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Clinical Trial to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of DA-4505 as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DA4505_AMST_I/IIa
Record Dates: First submitted 2024-02-15; First posted 2024-03-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monotherapy (Experimental): Phase 1a: Dose escalation Phase 1b: Dose expansion Phase 2a: Pharmacodynamic Biomarkers
  Interventions: Drug: DA-4505
- Combination with Pembrolizumab (Experimental): Phase 1a: Dose escalation Phase 1b: Dose expansion Phase 2a: Proof of concept Phase 2a: Pharmacodynamic Biomarkers
  Interventions: Drug: DA-4505 + Pembrolizumab

INTERVENTIONS:
Drug: DA-4505 — Phase 1a: Dose escalation Phase 1b: OBD and MTD Phase 2a: RP2D
  Arms: Monotherapy
Drug: DA-4505 + Pembrolizumab — Phase 1a/b: OBD, MTD of DA-4505 + 200mg of Pembrolizumab Phase 2a: RP2D of DA-4505 + 200mg of Pembrolizumab
  Arms: Combination with Pembrolizumab

SUMMARY:
This study is an Open-Label, Phase 1/2a, First-in-Human, Dose-Escalation, Dose-Expansion, and Proof-of-Concept Study to Investigate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of DA-4505 as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Locally Advanced or Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and older.
2. Capable of giving signed informed consent.
3. Diagnosed with particular disease characteristics.
4. Expected survival ≥ 3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
6. A female patient is eligible to participate if she is not pregnant or breastfeeding.
7. A male patient is eligible to participate if he agrees to remain abstinent or use a male condom when having sexual intercourse with a WOCBP, or if he has had a bilateral vasectomy.
8. Have measurable disease by revised RECIST v1.1 criteria.

Exclusion Criteria:

1. Inability to take oral medications or gastrointestinal abnormalities potentially impacting absorption.
2. Current enrollment or past participation in another clinical trial.
3. Unresolved adverse reactions (except alopecia) from previous cancer-directed therapy.
4. Use of cancer-directed therapies, including chimeric antigen receptor T cell therapy.
5. Autologous transplantation within 60 days.
6. Prior allogeneic transplantation.
7. Major surgery within 30 days, or unresolved complications after a major or minor surgery.
8. History of or currently active cardiovascular disease.
9. Clinically significant respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders.
10. History of other malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of adverse events (AEs) meeting protocol-defined dose-limiting toxicity(DLT) criteria | Cycle 1(21 days) in dose escalation
  The recommended Phase 2 dose(RP2D) will be the optimal biological dose (OBD) based on consideration of safety and tolerability information along with all available pharmacokinetic (PK), pharmacodynamic (PD), and efficacy data.
PK parameters for DA-4505 (Peak Plasma Concentration (Cmax)) | Day 1 and 2 of first 2 cycles (every 21 days)
  Determine DA-4505 Cmax
PK parameters for DA-4505 (Area Under the Curve (AUC)) | Day 1 and 2 of first 2 cycles (every 21 days)
  Determine DA-4505 AUC
PK parameters for DA-4505 (half-life (t1/2)) | Day 1 and 2 of first 2 cycles (every 21 days)
  Determine DA-4505 half-life (t1/2).
Response per revised "Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1) | approximately 12 months
  To determine the anti-tumor activity of both DA-4505 as a single agent and in combination with pembrolizumab

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul
  - Severance Hospital, Seoul